CLINICAL TRIAL: NCT01950871
Title: Diagnostic Performance of Prostate HistoScanningTM (PHS) in Men at Risk of Prostate Cancer Scheduled for an Initial Prostate Biopsy
Brief Title: Prostate Guided Biopsy Study Evaluating the Diagnostic Performance of Prostate HistoScanning
Acronym: PHSTT-01
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor is bankrupt
Sponsor: Advanced Medical Diagnostics s.a. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CR2P01127; DRKS00005263 (Registry Identifier: Deutsches Register Klinischer Studien)
Record Dates: First submitted 2013-09-19; First posted 2013-09-26 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2015-01

CONDITIONS: Prostate Cancer
Keywords: HistoScanning; TRUS; Prostate cancer; Biopsy guidance
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single arm study (Other): Prostate HistoScanning (HS) analysis with HS-guided biopsy will be used to sample two cores per suspicious area (displayed as red on an imaging monitor), up to a maximum of 3 suspicious areas per subject. Depending on the number of suspicious areas identified by prostate HS, the number of cores will be zero (if no suspicious area is identified) up to a maximum of 6 cores.
  Interventions: Device: Prostate HistoScanning

INTERVENTIONS:
Device: Prostate HistoScanning — In a single visit, subjects will first be imaged with TRUS for the purpose of generating data for prostate HS analysis. The results of HS analysis will be used later in the procedure. Subjects will then undergo two consecutive biopsy procedures. First, using TRUS, a systematic 10- to 12-core biopsy procedure will be performed. In turn, prostate HS data taken at the beginning of the procedure will be used to determine suspicious areas (displayed as red on an imaging monitor) and used to guide the biopsy procedure. Areas that are identified as suspicious (zero to a maximum of 3 areas) will then be sampled with two biopsy cores. Depending on the number of suspicious areas identified by prostate HS, the number of cores will be zero to a maximum of 6 cores.
  Other Names: PHS/PHS TT

SUMMARY:
The primary objective of the PHSTT-01 trial is to determine if prostate HistoScanning (HS) analysis can be used to improve the detection of clinically significant prostate cancer (PCa), and potentially reduce the burden and number of biopsies in routine clinical practice. Prostate HS is an ultrasound-based tissue characterization technology specifically developed to detect, visualize, and locate tissue suspected of harboring PCa. These suspicious tissues are displayed as red areas on an imaging monitor. Recently a new biopsy guidance tool has been developed that uses the results of the prostate HS analysis.

The subjects that will participate in this study are all scheduled for a first biopsy of the prostate. They will initially be imaged using transrectal ultrasound (TRUS) to obtain data for prostate HS analysis. The results of HS analysis will be used later in the procedure. Subjects will then undergo a routine systematic 10- to 12-core biopsy procedure using TRUS. This will be followed by a TRUS-guided biopsy that uses the result of prostate HS analysis and new biopsy guidance tool.

DETAILED DESCRIPTION:
PHSTT-01 is a multi-center, prospective clinical trial to evaluate the diagnostic performance of prostate HistoScanning (HS) analysis in men at risk of PCa that have been scheduled for a first prostate biopsy. The purpose of this study is to determine if prostate HS analysis can improve the detection of clinically significant PCa, and potentially reduce the burden and number of biopsies in routine clinical practice. Subjects are men with serum total prostate-specific antigen (PCA) <= 20ng/mL (<= 10ng/mL if taking the 5-alpha reductase inhibitor).

In a single visit, subjects will first be imaged with TRUS for the purpose of generating data for prostate HS analysis. The results of HS analysis will be used later in the procedure. Subjects will then undergo two consecutive biopsy procedures. First, using TRUS, a systematic 10- to 12-core biopsy procedure will be performed. In turn, prostate HS data taken at the beginning of the procedure will be used to determine suspicious areas (displayed as red on an imaging monitor) and used to guide the biopsy procedure. Areas that are identified as suspicious (zero to a maximum of 3 areas) will then be sampled with two biopsy cores. Depending on the number of suspicious areas identified by prostate HS, the number of cores will be zero to a maximum of 6 cores.

ELIGIBILITY:
Inclusion Criteria:

* Men at risk of PCa scheduled for first biopsy with serum total PSA

  ≤ 20 ng/ml (≤ 10 ng/mL if taking 5-alpha reductase inhibitors) from maximally 3 months ago
* Signed informed consent

Exclusion Criteria:

* Previous prostate biopsy
* Confirmed PCa
* PSA > 20 ng/ml (or > 10 ng/mL if taking 5-alpha reductase inhibitors)
* Active urinary tract infection
* Presence/history of any confirmed cancer
* Recent prostatic surgery (past 6 months)
* History of pelvic radiotherapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance of prostate HistoScanning (HS) to identify clinically significant PCa using histology outcomes from systematic prostate biopsy (Bx) as reference | 1 year
  Compare prostate HS results to the systematic Bx outcome (positive or negative) for clinically significant PCa (defined as Gleason sum ≥ 7) in the non-run-in population.

SECONDARY OUTCOMES:
Diagnostic performance of prostate HS to identify PCa using histology outcomes from systematic Bx as reference | 1 year
  Compare prostate HS results to the systematic Bx outcome (positive or negative) for all PCa in the non-run-in population.
Diagnostic performance of prostate HS to identify clinically significant PCa using a combination of outcomes of both systematic Bx and HS-guided biopsy histology as reference | 1 year
  Compare prostate HS results to the combination of systematic and HS-guided Bx outcomes (positive or negative) for clinically significant PCa (defined as Gleason sum ≥ 7) in the non-run-in population.
Difference in detection rates of clinically significant PCa between systematic and HS-guided biopsy. | 1 year
  Compared PCa detection rates of systematic and HS-guided prostate Bx in the non-run-in population.

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Tombal, Prof, Principal Investigator — Cliniques Universitaires Saint-Luc, Brussels, Belgium
Locations (34):
- Austria (3):
  - Krankenhaus der Barmherzigen Brüder, Vienna
  - Medical Center Hanuschkrankenhaus, Vienna
  - Medical Center Med.Landeskrankenhaus Vöcklabruck, Vöcklabruck
- Belgium (3):
  - University Medical Center UZ VUB, Brussels, Brussels Capital
  - • University Medical Center Cliniques Universitaires Saint Luc, Brussels, Brussels Capital
  - Medical Center Onze Lieve Vrouw Ziekenhuis OLVZ, Aalst
- University Medical Center St. Marina University Hospital, Varna, Bulgaria
- Czechia (2):
  - Medical Center Urologická klinika - Fakultní nemocnice, Olomouc
  - University Medical Center Všeobecná fakultní nemocnice v Praze (VFN) a 1. -General University Hospital and First Faculty of Medicine Charles University, Prague
- • University Medical Center Urinary Tract Surgery - Urology Dpt - Odense Universitetshospital Svendborg Sygehus, Odense C, Denmark
- Medical Center North-Estonian Medical Center Foundation, Tallinn, Estonia
- France (2):
  - Medical Center Institut Mutualiste Montouris, Paris
  - University Medical Center CHU Saint Etienne, Saint-Etienne
- Germany (8):
  - Medical Center Cancer Center - Prostatazentrum, Braunschweig
  - Medical Center PAN Klinik, Cologne
  - Medical Center Paracelsus Klinik, Düsseldorf
  - Medical Center Martini Klinik - Prostate Cancer Center, Hamburg
  - Medical Center Klinikum Herford, Herford
  - Medical Center St. Elisabeth Krankenhaus, Leipzig
  - Medical Center Klinikum Leverkusen, Leverkusen
  - Medical Center Klinikum Wolfsburg Urologie, Wolfsburg
- Medical Center Uro-Clin Ltd, Pécs, Hungary
- University Medical Center University Vita-Salute, Scientific Institute H. San Raffaele, Milan, Italy
- Medical Center URO, Riga, Latvia
- University Medical Center Vilniaus Universiteto Onkologijos Institutas - Santariškiu Clinics, Vilnius, Lithuania
- Medical Center Antoni Van Leeuwenhoek Ziekenhuis - Nederlands Kanker Instituut, Amsterdam, Netherlands
- University Medical Center Moscow State University of Medicine and Dentistry named after A.I.Evdokimov, Moscow, Russia
- University Medical Center Vall d'Hebron University Hospital - Autonoma Universitat Barcelona, Barcelona, Spain
- Carouge medical centre, Carouge, Switzerland
- Turkey (Türkiye) (2):
  - Medical Center URO-TIP Urological Diagnosis Center, Istanbul
  - Medical Center Acıbadem Kozyatağı Hospital, Istanbul
- United Kingdom (3):
  - Medical Center Blackpool Victoria Hospital, Blackpool
  - University Medical Center Nuffield Health - University Hospitals Bristol (UHB) - Bristol Royal Infirmary and Southmead Hospitals, Bristol
  - Medical Center Spire Washington Hospital, Tyne and Wear